CLINICAL TRIAL: NCT05635851
Title: NO AD: Use of Nitric Oxide (NO) Donors for the Prevention of Autonomic Dysreflexia (AD) During Bowel Care Following SCI
Acronym: NO AD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Dr. Victoria Claydon, Professor, Principal Investigator, Simon Fraser University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H22-00878
Record Dates: First submitted 2022-10-04; First posted 2022-12-02 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Spinal Cord Injuries; Autonomic Dysreflexia
Keywords: spinal cord injury; autonomic dysreflexia; blood pressure; bowel care management; defecation
MeSH Terms: conditions — Spinal Cord Injuries; Autonomic Dysreflexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glyceryl trinitrate sublingual spray (Experimental): Glyceryl trinitrate (GTN) sublingual spray will be administered up to three times every fifteen minutes, each dose being 0.4mg.
  Interventions: Drug: Glyceryl Trinitrate Only Product in Oromucosal Dose Form
- Placebo sublingual spray (Placebo Comparator): An approximate flavour-matched placebo sublingual spray will be administered up to three times every fifteen minutes.
  Interventions: Other: Placebo sublingual spray

INTERVENTIONS:
Drug: Glyceryl Trinitrate Only Product in Oromucosal Dose Form — Glyceryl trinitrate will be administered via sublingual spray.
  Other Names: GTN
  Arms: Glyceryl trinitrate sublingual spray
Other: Placebo sublingual spray — A placebo sublingual spray will be administered.
  Other Names: Placebo spray
  Arms: Placebo sublingual spray

SUMMARY:
This project aims to evaluate the safety and efficacy of using a short-acting drug to reduce the maximal blood pressure during dangerous blood pressure spikes that happen during bowel care in individuals with spinal cord injury. the investigators will monitor the physiological effects of this drug during at-home bowel care to best understand the drug's effects in typical use.

DETAILED DESCRIPTION:
Purpose: The primary purpose of this study is to investigate the effects of sublingual nitric oxide (NO) donor spray on cardiovascular changes triggered by bowel care.

Hypothesis: NO donor spray will lower the maximum blood pressure spikes during high blood pressure events triggered by bowel care in people with spinal cord injury.

Justification: In people with spinal cord injury, episodes of high blood pressure are common during strong sensory stimuli such as those present during routine bowel care. These episodes of high blood pressure can be dangerous due to the magnitude of blood pressure increase and because they can be accompanied by irregular heart beats. This condition, known as autonomic dysreflexia (AD), is most common in individuals with high-level injuries.

The experience of autonomic dysreflexia can vary widely between individuals: some have goosebumps, sweating, facial flushing or headaches, while others have no symptoms at all, despite their changes in heart rate and blood pressure.

One possible approach to help manage AD is the use of fast-acting, short-term vasodilators such as nitric oxide (NO) donors (e.g. glyceryl trinitrate, GTN) to decrease blood pressure during AD experienced during bowel care. This approach is already part of the clinical recommendations for management of AD during bowel care, and yet its safety and efficacy have never been tested during at-home bowel care. Currently, a sublingual GTN spray is not often used in the home setting, although it is thought that using this medication might reduce the cardiovascular effects of bowel care after spinal cord injury. The long-term consequences of these short-term elevations in blood pressure during autonomic dysreflexia are not fully understood, but given that they are often associated with discomfort, and have been known to be associated with more severe events such as stroke, it would be beneficial to reduce their occurrence during daily care routines.

Objectives: The investigators aim to evaluate whether GTN improves AD during normal at-home bowel care.

Research Design: The study is a randomised placebo-controlled double-blind crossover clinical trial to evaluate the effect of sublingual GTN (spray) on beat-to-beat cardiovascular responses to normal bowel care in 26 individuals with chronic high-level SCI who are known to have AD.

Statistical Analysis: Data will be analysed using R statistical software. Mean maximum blood pressure and mean drop in systolic blood pressure will be calculated. Mean time to onset of drug action will also be calculated. A paired t-test will be used to determine if there is a significant within-participant difference in the change of mean maximum blood pressure values or mean drop in systolic blood pressure between the placebo and the GTN conditions. Two-way repeated measures ANOVA will be used to compare symptoms, test conditions, and test phases. Categorical data will be analysed with Spearman's rank correlations and linear regressions to determine if any findings correlate with biological variables including level of injury, sex, and cardiovascular variables.

ELIGIBILITY:
Inclusion Criteria:

* participants must have had a traumatic spinal cord injury at least one year ago
* regular bowel care routine
* can communicate in English

Exclusion Criteria:

* cauda equina or conus lesions
* currently use ventilator
* colostomy, or do not perform regular bowel care
* skin breakdown (pressure sores)
* cannot communicate in English
* under 19 years old
* possibly or certainly pregnant
* medical/psychiatric condition or substance abuse that is likely to affect ability to complete study
* currently using medications containing PDE-5 inhibitors
* currently using medications containing GTN
* allergy to GTN

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Blood pressure change during bowel care | Time Frame: Measured continuously during bowel care (approximately one hour) on two occasions within 28 days.
  Beat-to-beat blood pressure will be recorded using a finger blood pressure cuff (Finometer) on two occasions within 28 days, for up to one hour on each occasion.

SECONDARY OUTCOMES:
Change in symptoms of autonomic dysreflexia | Time Frame: Measured upon completion of bowel care (approximately one hour) on two occasions within 28 days.
  Symptoms will be recorded after each arm of testing to determine if the drug condition improves symptoms
Incidence of arrhythmia | Time Frame: Measured continuously during bowel care (approximately one hour) on two occasions within 28 days.
  Beat-to-beat ECG will be recorded using a Finometer on two occasions within 28 days, for up to one hour on each occasion.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Claydon, PhD, Principal Investigator — Simon Fraser University